CLINICAL TRIAL: NCT02324179
Title: Use of EndoPAT for Measurements of Endothelial Dysfunction in HIV Infected Children and Healthy Controls
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Grace McComsey, Grace McComsey, MD, FIDSA, University Hospitals Cleveland Medical Center
Other Study IDs: 05-14-22; 05-14-22 (Other: University Hospital IRB)
Record Dates: First submitted 2014-08-28; First posted 2014-12-24 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: HIV; Endothelial Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive: people with HIV diagnosis
- Control (HIV negative): people without HIV

SUMMARY:
Our objective is to determine whether HIV infected youth have higher level of endothelial dysfunction, as measured by Peripheral Arterial Tonometry, when compared to age matched healthy controls. The investigators also aim to gather preliminary data on whether endothelial Peripheral Arterial Tonometry (endoPAT) measurements of endothelial dysfunction are independently associated with HIV and antiretroviral factors, and with markers of inflammation and traditional cardiovascular disease risk.

DETAILED DESCRIPTION:
Study Objectives and Hypothesis Our objective is to determine whether HIV infected youth have higher level of endothelial dysfunction, as measured by Peripheral Arterial Tonometry, when compared to age matched healthy controls. We also aim to gather preliminary data on whether endoPAT measurements of endothelial dysfunction are independently associated with HIV and antiretroviral factors, and with markers of inflammation and traditional cardiovascular disease risk.

Specific Aim 1:

To compare endothelial function, as measured by endoPAT, between HIV-infected youth and matched healthy controls.

Hypothesis: HIV infected youths will have impaired endothelial function compared to age matched healthy controls.

Specific Aim 2:

To determine risk factors of endothelial dysfunction by evaluating: 1) risk factors specific to HIV such as disease stage, cluster of differentiation 4 (CD4) count, HIV viral load, specific ART regimen, perinatally acquired versus behaviorally acquired infection; 2) markers of cardiovascular disease risk such as smoking, lipid levels, insulin resistance; 3) markers of inflammation and immune activation Hypothesis: Endothelial dysfunction will correlate with advanced HIV disease stage, use of protease inhibitors and worse traditional cardiovascular disease risk factors including lipids, insulin resistance, and smoking.

Specific Aim 3:

To assess whether endothelial function changes over a period of 24 weeks in HIV infected youths and controls.

Hypothesis: Endothelial dysfunction will progress over time in HIV-infected children but not in healthy controls.

Study Design This is a 24-week observational cohort study to gather preliminary data on the prevalence and risk factors for endothelial dysfunction in HIV-infected youths. Children enrolled will be between the ages of 8 and 30 years and either congenitally or behaviorally infected with HIV, on continuous ART for at least 6 months and with HIV-1 RNA <1,000 copies/mL. We will also enroll an age- and gender-matched group of healthy controls. A total of 50 HIV-infected children/young adults and 50 matched controls will be enrolled.

Evaluations will be performed at two time points: baseline and week 24. At both visits, evaluations will be similar. We will collect demographic data and medical history including date of birth, sex, gender, CD4 cell count nadir, past and current ART and non-ART medication history, HIV stage based on the CDC guidelines, HIV diagnosis date and method of HIV acquisition, alcohol, smoking and drug habits, as well as family history of cardiovascular disease or diabetes. We will record clinical measurements including blood pressure, physical examination abnormalities, waist and hip circumferences and tanner stage. Subjects will undergo laboratory measurements of lipids levels and markers of insulin resistance in a fasting state (>8 hrs fast except for water and medications), as well as inflammation and immune activation markers (hsCRP, Interleukin 6 or IL-6, sCD14). HIV RNA and CD4 cell count will be collected from clinical records. Plasma and serum will be stored for possible future measurements of other inflammation and cardiovascular markers. We will perform endothelial function measurements by PAT as recommended by the manufacturer.

Controls will be recruited from the community using Institutional Review Board (IRB)-approved flyers, as uninfected siblings or relatives of the HIV-infected patients, or from physician referrals.

ELIGIBILITY:
Inclusion Criteria:

* For HIV+ group:
* age 8-30 years of age
* HIV infection
* On continuous ART for at least 6 months
* HIV-1 RNA < 1,000 copies/mL performed in the past 5 months

For healthy controls:

* age and gender matched 1:1 to HIV-positive subjects
* absence of known HIV or other medical conditions that may affect systemic inflammation
* Not receiving or prescribed any regular chronic medications.

Exclusion Criteria:

* - Active illness or regular medication
* Diabetes
* Known coronary artery disease
* Pregnancy and or lactation

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. HIv positive: subjects seen at the Special Immunology Unit
  2. Controls: HIV-negative controls will be healthy people who are friends or family members of the HIV-infected patients, or employees who are not employed by the principal investigator or the co-investigators or recruited through researchmatch.org
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
endothelial function, as measured by endoPAT, between HIV-infected youth and matched healthy controls | one year
  Endothelial function will be measured using peripheral arterial tonometry. The device will record finger arterial pulsatile volume changes. The recordings will be performed with the patient in supine position with both hands at the same level. A blood pressure cuff will be placed on the upper arm (non-dominant); the probes will be placed on the finger of each hand (same finger on both hands) and continuing recording of blood volume responses from both hands will be initiated. After a period of stabilization, the blood pressure cuff on the study arm will be inflated to 60 mm Hg above systolic pressure for 5 min. The cuff will be deflated to induce reactive hyperemia and assess PAT. A reactive hyperemia index will be generated and is the post to pre occlusion PAT signal ratio in the occluded side normalized to the control side and corrected for baseline vascular tone. A normal index is >1.67 and abnormal is ≤ 1.67.
risk factors of endothelial dysfunction | one year
  To determine risk factors of endothelial dysfunction by evaluating: 1) risk factors specific to HIV such as disease stage, CD4 count, HIV viral load, specific ART regimen, perinatally acquired versus behaviorally acquired infection; 2) markers of cardiovascular disease risk such as smoking, lipid levels, insulin resistance; 3) markers of inflammation and immune activation
endothelial function changes over a period of 24 weeks in HIV infected youths and controls. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Special Immunology Unit, Cleveland, Ohio, United States

REFERENCES:
- [Result] Bonetti PO, Barsness GW, Keelan PC, Schnell TI, Pumper GM, Kuvin JT, Schnall RP, Holmes DR, Higano ST, Lerman A. Enhanced external counterpulsation improves endothelial function in patients with symptomatic coronary artery disease. J Am Coll Cardiol. 2003 May 21;41(10):1761-8. doi: 10.1016/s0735-1097(03)00329-2. PMID 12767662
- [Result] Escarcega RO, Franco JJ, Mani BC, Vyas A, Tedaldi EM, Bove AA. Cardiovascular disease in patients with chronic human immunodeficiency virus infection. Int J Cardiol. 2014 Jul 15;175(1):1-7. doi: 10.1016/j.ijcard.2014.04.155. Epub 2014 Apr 21. PMID 24798779
- [Result] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Nedeljkovic ZS, Menzoian JO, Vita JA. Predictive value of noninvasively determined endothelial dysfunction for long-term cardiovascular events in patients with peripheral vascular disease. J Am Coll Cardiol. 2003 May 21;41(10):1769-75. doi: 10.1016/s0735-1097(03)00333-4. PMID 12767663
- [Result] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169
- [Result] Hamburg NM, Palmisano J, Larson MG, Sullivan LM, Lehman BT, Vasan RS, Levy D, Mitchell GF, Vita JA, Benjamin EJ. Relation of brachial and digital measures of vascular function in the community: the Framingham heart study. Hypertension. 2011 Mar;57(3):390-6. doi: 10.1161/HYPERTENSIONAHA.110.160812. Epub 2011 Jan 24. PMID 21263120
- [Result] Hijmering ML, Stroes ES, Pasterkamp G, Sierevogel M, Banga JD, Rabelink TJ. Variability of flow mediated dilation: consequences for clinical application. Atherosclerosis. 2001 Aug;157(2):369-73. doi: 10.1016/s0021-9150(00)00748-6. PMID 11472736
- [Result] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Result] Moerland M, Kales AJ, Schrier L, van Dongen MG, Bradnock D, Burggraaf J. Evaluation of the EndoPAT as a Tool to Assess Endothelial Function. Int J Vasc Med. 2012;2012:904141. doi: 10.1155/2012/904141. Epub 2012 Feb 14. PMID 22500237
- [Result] Poredos P. Endothelial dysfunction in the pathogenesis of atherosclerosis. Int Angiol. 2002 Jun;21(2):109-16. PMID 12110769
- [Result] Poredos P, Jezovnik MK. Testing endothelial function and its clinical relevance. J Atheroscler Thromb. 2013;20(1):1-8. doi: 10.5551/jat.14340. Epub 2012 Sep 10. PMID 22972428
- [Result] Schnabel RB, Schulz A, Wild PS, Sinning CR, Wilde S, Eleftheriadis M, Herkenhoff S, Zeller T, Lubos E, Lackner KJ, Warnholtz A, Gori T, Blankenberg S, Munzel T. Noninvasive vascular function measurement in the community: cross-sectional relations and comparison of methods. Circ Cardiovasc Imaging. 2011 Jul;4(4):371-80. doi: 10.1161/CIRCIMAGING.110.961557. Epub 2011 May 6. PMID 21551420
- [Result] Schnall RP, Shlitner A, Sheffy J, Kedar R, Lavie P. Periodic, profound peripheral vasoconstriction--a new marker of obstructive sleep apnea. Sleep. 1999 Nov 1;22(7):939-46. PMID 10566912
- [Result] Selamet Tierney ES, Newburger JW, Gauvreau K, Geva J, Coogan E, Colan SD, de Ferranti SD. Endothelial pulse amplitude testing: feasibility and reproducibility in adolescents. J Pediatr. 2009 Jun;154(6):901-5. doi: 10.1016/j.jpeds.2008.12.028. Epub 2009 Feb 12. PMID 19217124
- [Result] Widlansky ME, Gokce N, Keaney JF Jr, Vita JA. The clinical implications of endothelial dysfunction. J Am Coll Cardiol. 2003 Oct 1;42(7):1149-60. doi: 10.1016/s0735-1097(03)00994-x. PMID 14522472
- [Result] Xu Y, Arora RC, Hiebert BM, Lerner B, Szwajcer A, McDonald K, Rigatto C, Komenda P, Sood MM, Tangri N. Non-invasive endothelial function testing and the risk of adverse outcomes: a systematic review and meta-analysis. Eur Heart J Cardiovasc Imaging. 2014 Jul;15(7):736-46. doi: 10.1093/ehjci/jet256. Epub 2014 Jan 7. PMID 24399339
- [Result] Antiretroviral Therapy Cohort Collaboration. Causes of death in HIV-1-infected patients treated with antiretroviral therapy, 1996-2006: collaborative analysis of 13 HIV cohort studies. Clin Infect Dis. 2010 May 15;50(10):1387-96. doi: 10.1086/652283. PMID 20380565